CLINICAL TRIAL: NCT03360266
Title: Comparative Evaluation of Remineralizing Efficacy of Fluoride Varnish and Its Combination Varnishes on White Spot Lesions in Children With ECC: A Randomized Clinical Trial
Brief Title: Evaluation of Remineralizing Efficacy of Combination Varnishes on White Spot Lesions in ECC Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indira Gandhi Institute of Dental Science (Other)
Responsible Party: Principal Investigator, DR.S.RADHA, Principal investigator, Indira Gandhi Institute of Dental Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIGIDSIIRB2015 NDP20PGRSPPD
Record Dates: First submitted 2017-10-30; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Child; Early Childhood Caries
Keywords: remineralization; fluoride varnish
MeSH Terms: interventions — Sodium Fluoride; Enamel Pro Varnish

STUDY DESIGN:
Intervention Model Description: The study model involves three groups
Who Masked: Investigator
Masking Description: Investigator is masked in application of fluoride varnish and during all followup visits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Profluorid group (Active Comparator): 5% Sodium Fluoride varnish (Profluorid varnish) applied over white spot lesions on maxillary anterior teeth
  Interventions: Combination Product: Sodium Fluoride with CPP-ACP varnish; Combination Product: sodium fluoride with ACP varnish
- Enamel Pro (Experimental): Sodium Fluoride with ACP varnish (Enamel Pro varnish) applied over white spot lesions on maxillary anterior teeth
  Interventions: Combination Product: Sodium Fluoride with CPP-ACP varnish; Drug: 5% Sodium Fluoride Varnish
- MI varnish (Experimental): Sodium Fluoride with CPP-ACP varnish (MI varnish) applied over white spot lesions on maxillary anterior teeth
  Interventions: Combination Product: sodium fluoride with ACP varnish; Drug: 5% Sodium Fluoride Varnish

INTERVENTIONS:
Combination Product: Sodium Fluoride with CPP-ACP varnish — for children with ECC, this varnish effectively remineralizes the white spot lesion
  Other Names: MI varnish
  Arms: Enamel Pro; Profluorid group
Combination Product: sodium fluoride with ACP varnish — for children with ECC, this varnish effectively remineralizes the white spot lesion
  Other Names: Enamel Pro
  Arms: MI varnish; Profluorid group
Drug: 5% Sodium Fluoride Varnish — ffor children with ECC, this varnish effectively remineralizes the white spot lesion
  Other Names: Profluorid
  Arms: Enamel Pro; MI varnish

SUMMARY:
The remineralizing efficacy of 3 fluoride varnishes were assessed in children with white spot lesion under 6 years of age ( children with early childhood caries)

DETAILED DESCRIPTION:
Early childhood caries (ECC) is the presence of 1 or more decayed (Non - Cavitated or Cavitated lesions), missing (due to caries) or filled tooth surface in any primary tooth in a child of 71 months of age or younger. In children younger than 3 years of age, any sign of smooth-surface caries is indicative of severe early childhood caries (S-ECC). It is a virulent form of caries, which develops on smooth surfaces and progresses rapidly. In children aged 12 to 30 months it initially affects the maxillary primary incisors and first primary molars, reflecting the pattern of eruption.

In ECC, the first clinical observation of demineralization in enamel is the white spot lesion, which is characterized by enamel demineralization of the subsurface, with increasing porosity due to the removal of minerals into the outer surface. At this stage, the caries lesion is usually reversible.

In young children, remineralization can be achieved by Non- invasive methods that are very effective. Fluoride prevents the caries process, leading to the formation of less soluble fluorapatite crystals. Among them, Topical fluorides are the most respected regimen. On application of topical fluorides to the teeth, calcium fluoride-like globules are formed on the tooth surface. These globules are effective mineral reservoirs that help prevent demineralization and promote remineralization by releasing calcium, phosphate and fluoride following acid attacks.

American Academy of Pediatric Dentistry (AAPD) recommends fluoride varnish in children. Randomized control trials have found it to be efficacious in primary teeth. Fluoride varnish can reverse or arrest caries lesions as well as prevent demineralization process of an incipient caries/white spot lesion, when combined with other preventive measures such as oral hygiene instructions & diet counseling.Children at increased caries risk should receive a professional fluoride treatment at least every six months. There is evidence from randomized controlled trials and meta-analyses that professionally applied topical fluoride treatments as five percent sodium fluoride varnish or 1.23 percent fluoride gel preparations are efficacious in reducing caries in children at caries risk.

Fluoride varnish works by increasing the concentration of fluoride in the outer surface of teeth, thereby enhancing fluoride uptake during early stages of demineralization. The varnish hardens on the tooth as soon as it contacts saliva, allowing the high concentration of fluoride to be in contact with tooth enamel for an extended period of time This is a much longer exposure compared to other high-dose topical fluorides such as gels or foams, with less risk of fluorosis even in children younger than 6 years.

It has been observed from the literature review that only invitro studies and few clinical studies have been done in treating WSL in orthodontic patients using these combination varnishes. To our Knowledge, no clinical studies has assessed its efficacy and compared the effectiveness of these combination varnishes in remineralising white spot lesions of ECC in young children. Thus, this study was planned to compare the remineralizing efficiency of fluoride varnish with a combination of fluoride and calcium phosphate varnishes on white spot lesions in smooth surfaces of primary anterior teeth of children with ECC.

ELIGIBILITY:
Inclusion Criteria:

1. Preschool children with ECC.
2. Children with active white spot lesions on labial surface of 1 or more primary maxillary anterior teeth.
3. Children whose parents signed the informed consent form/willing to participate in the study.
4. Apart from fluoride varnish and fluoridated tooth paste, subjects exposed to no other form of fluoride were included.

Exclusion Criteria:

1. Preschool children with cavitated lesions on primary maxillary anterior teeth.
2. Developmental enamel alterations (hypoplasia, fluorosis).
3. Children with systemic diseases.
4. Children with allergy to milk products.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2016-12-24 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Dimension and Activity of white spot lesions. | 6 months
  The dimension of white spot lesions were measured with photographs using Adobe photoshop software. After prolonged air drying of 5 sec, the activity of white spot lesions were visualized using CPITN probe

CONTACTS AND LOCATIONS:
Overall Officials: Kayalvizhi Gurusamy, MDS, Study Director — IGIDS

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radha S, Kayalvizhi G, Adimoulame S, Prathima GS, Muthusamy K, Ezhumalai G, Jagadesaan N. Comparative Evaluation of the Remineralizing Efficacy of Fluoride Varnish and its Combination Varnishes on White Spot Lesions in Children with ECC: A Randomized Clinical Trial. Int J Clin Pediatr Dent. 2020 Jul-Aug;13(4):311-317. doi: 10.5005/jp-journals-10005-1673. PMID 33149400